CLINICAL TRIAL: NCT02215018
Title: Safety, Tolerability and Pharmacokinetics of BI 44370 TA Oral Drinking Solution in Healthy Male Volunteers (Dose Range: 5 - 800 mg). A Double-blind (Within Dose Groups), Randomised, Placebo-controlled Within Dose Groups, Single Rising Dose Study, Including Re-dosing at 100 mg and 500 mg (Solution) and at 200 mg (Four 50 mg Tablets)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 44370 TA Oral Drinking Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1246.1
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (4):
- BI 44370 TA solution (Experimental)
  Interventions: Drug: BI 44370 TA solution
- BI 44370 TA tablet (Experimental)
  Interventions: Drug: BI 44370 TA tablet
- Placebo solution (Placebo Comparator)
  Interventions: Drug: Placebo solution
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: BI 44370 TA solution
  Arms: BI 44370 TA solution
Drug: BI 44370 TA tablet
  Arms: BI 44370 TA tablet
Drug: Placebo solution
  Arms: Placebo solution
Drug: Placebo tablet
  Arms: Placebo tablet

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics of single rising oral doses of BI 44370 TA in healthy male volunteers, to compare a drinking solution vs. a tablet formulation and to assess intra-individual pharmacokinetic (PK) variability by re-dosing two further doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR, RR and body temperature), 12-lead ECG, clinical laboratory tests
2. Age ≥21 and Age ≤50 years
3. Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR), Respiratory rate (RR) , body temperature and Electrocardiogram(ECG)) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
21. A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
22. Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 10 days after last drug administration
Number of patients with clinically significant findings in vital signs | up to 10 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 10 days after last drug administration
Number of patients with clinically significant findings in ECG | up to 10 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 10 days after last drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 72 hours after drug administration
tz (time of last measurable concentration of the analyte in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTp.o. (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase tz following an extravascular dose) | up to 72 hours after drug administration
λz (the terminal rate constant) | up to 72 hours after drug administration
Aet1/t2 (total quantity of analyte excreted in the urine in the time interval from t1 to t2) | up to 24 hours after drug administration
fet1/t2 (the fractional excretion of the analyte in the time interval from t1 to t2) | up to 24 hours after drug administration
CLR,t1/t2 (the renal clearance of the analyte in the time interval from t1 to t2) | up to 24 hours after drug administration